CLINICAL TRIAL: NCT00203216
Title: A Single-Center, Open-Label Trial Examining the Efficacy and Safety of Levetiracetam for the Prophylactic Treatment of Migraine, With or Without Aura
Brief Title: A Clinical Study Examining the Safety and Effectiveness of a New Medication (Keppra®) for the Prevention of Migraine Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: William B. Young, M.D.-Principal Investigator, Thomas Jefferson University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WBY/LEV01; 080-19000-H80001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Levetiracetam; Transcranial Magnetic Stimulation

ARMS (1):
- Levatiracetam (Experimental): Subject titrated open-label study drug to maximally tolerated dose: maximum: 3000 mg. per date. (minimum allowed daily dose to remain in study: 1000)
  Interventions: Drug: levetiracetam; Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Drug: levetiracetam — Daily dose of open label levatiracetam was 3000 mg. or maximally tolerated dose. (Maximum daily dose: 3000 mg. Minimum daily dose allowed for study participation:1000 mg)
  Other Names: Keppra
Procedure: Transcranial Magnetic Stimulation

SUMMARY:
The study drug levetiracetam is FDA approved as an add-on medication in the treatment of partial onset seizures in adults with epilepsy. The trade name is Keppra®. This is an "open-label" trial, which means that all participating patients will receive active study drug.

The Jefferson Headache Center has developed this clinical study to evaluate the safety and effectiveness of levetiracetam in preventing migraine headaches, with or without aura (visual disturbances).

In addition, the study site will be performing a procedure called Transcranial Magnetic Stimulation (TMS). This procedure measures brain activity because it is thought that people with migraine experience periods of cortical hyperexcitability or over-activity in the brain. This information may help physicians in the future determine which preventive medications will work for which patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between the ages of 18 and 65
* Patient has an IHS diagnosis of migraine with or without aura for at least one-year prior to screening
* Patient has experienced between 4 and 10 migraine headaches per month over the past six months, with at least 48 hours separating attacks
* Patient is able to differentiate migraine attacks from other headache types, if applicable
* Patient is not currently and has not in the 4 weeks preceding screening received prophylactic treatment for the indication of migraine
* Patients daily medications have remained at a stable dose for the 4 weeks preceding screening
* Patient is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female of child-bearing potential
* Patient has negative urine pregnancy test prior to study entry, if female of child-bearing potential
* Patient is able to understand and comply with all study requirements
* Patient provides written informed consent prior to any screening procedures being conducted

Exclusion Criteria:

* Women who are pregnant or lactating
* Patients with onset of migraine after 50 years of age
* Patients who experience > 15 headache days per month
* Patients who have been previously treated or are currently being treated with levitiracetam
* Patients who have failed greater than 3 adequate trials of other antiepileptic drugs for the prevention of migraine.
* Patients who, in the investigators opinion, have a history or have evidence of a medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial
* Patients with an abnormal ECG that, in the investigators opinion, would expose them to increased risk of adverse events or interfere with study drug and/or analysis of efficacy/tolerability
* Patients who take medication for acute treatment greater than 10 days per month over the past three months.
* Patients who are allergic to or have shown hypersensitivity to compounds similar to levetiracetam
* Patients with a history of significant drug or alcohol abuse within the past year
* Patients who have had a suicidal ideation in the 3 months prior to screening or has a history of attempted suicide
* Patients who currently have or have a history of significantly impaired renal function
* Patients who have participated in an investigational drug trial in the 30 days prior to the screening visit
* Patients who have a Beck Depression Inventory score of > 18 at screening
* Patients who have > 0 on question number 9 of Beck Depression Inventory (Suicidal Thoughts or Wishes question)
* Patients who have a defibrillator or pacemaker, an implanted medication pump, a metal plate in the skull, or metal objects inside the eye or skull (e.g. a shrapnel wound).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-09; Primary Completion 2005-01 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Young, MD, Principal Investigator — Thomas Jefferson University, Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Levetiracetam/Transcranial Magnetic Stimulation: In this open label trial, all subjects will receive levetiracetam. Subjects may be titrated up to their maximum tolerated dose (MTD) or 3000 mg daily, whichever is lowest. Subjects who cannot tolerate a dose of at least 1000mg per day will be discontinued from the trial. Transmagnetic stimulation will be performed to measure cortical excitability at various intervals during the study.
Period: Overall Study
Arm/Group | Levetiracetam/Transcranial Magnetic Stimulation
Started | 31
Completed | 27
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Levetiracetam/Transcranial Magnetic Stimulation
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is Defined as Average Change in Frequency of Migraine Attacks Over Each 4-week Interval of the Treatment Period as Compared to the 4-week Baseline Period.
Description: Number of migraine attacks will be measured at baseline (28 day period prior to start of study medication). The baseline number of attacks will be compared to that in the following 28 day intervals:
  * visit_4 = first follow-up interval (0 to 28 days after starting study drug)
  * visit_5 = second follow-up interval (28 to 56 days)
  * visit_6 = third follow-up interval (56 to 84 days)
  * visit_7 = fourth follow-up interval (84 to 126 days) The change in headache attacks post-treatment will be averaged in a multiple regression model, looking at the following: visit number, age, gender, BMI
Time Frame: Compare frequency of migraine attacks in baseline period to the average of the change following these 28 day periods prior to: Visit 4 (day 0-28), visit 5 (day 28-56), visit 6 (day 576-84), visit 7 (day 84-126).
Measure: Mean (Standard Deviation); unit: migraine attacks per month
Arm/Group | Levetiracetam/Transcranial Magnetic Stimulation
Number analyzed (Participants) | 31
migraine attacks per month | -0.058 (5.10)

2. Secondary Outcome: Change in Number of Migraine Days Over Each 4-week Interval of the Treatment Period as Compared to the 4-week Baseline Period
Description: Number of migraine attacks will be measured at baseline (28 day period prior to start of study medication). The baseline number of attacks will be compared to that in the following 28 day intervals:
  * visit_4 = first follow-up interval (0 to 28 days after starting study drug)
  * visit_5 = second follow-up interval (28 to 56 days)
  * visit_6 = third follow-up interval (56 to 84 days)
  * visit_7 = fourth follow-up interval (84 to 126 days)
Time Frame: Baseline period (day -28 to day 0) compared to the 28 day period prior to Visit 4-7.
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: migraine days

3. Secondary Outcome: Change in Average Severity if Migraine Attacks Per Each Consecutive 4-week Interval of the Treatment Period as Compared to the 4-week Baseline Period
Time Frame: Baseline period compared to 28 day interval prior to Visit 4-7.
Reporting Status: Not Posted
Measure: Median (Inter-Quartile Range); unit: severity rating

4. Secondary Outcome: Change in Use of Acute Agents Attacks Per Each Consecutive 4-week Interval of the Treatment Period as Compared to the 4-week Baseline Period.
Time Frame: Baseline period compared to the 28 day period prior to each of the following visits: Visit 4-7.
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: number of acute medications used

ADVERSE EVENTS:
Arm/Group | Levetiracetam/Transcranial Magnetic Stimulation
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 21/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam/Transcranial Magnetic Stimulation (N=31)
fatigue (Nervous system disorders) | 21 (21)
Irritability (Nervous system disorders) | 16 (16)
Dizziness (Nervous system disorders) | 13 (13)
Labile mood (Psychiatric disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes